CLINICAL TRIAL: NCT02862613
Title: Clinical Study Using Precision Cell Immunotherapy Combined With Transcatheter Arterial Chemoembolization in Advanced Liver Cancer
Brief Title: Precision Cell Immunotherapy Combined With TACE in Advanced Liver Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai International Medical Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIMC-20160106
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Precision Cells; Transcatheter Arterial Chemoembolization; Advanced Liver Cancer
Keywords: Precision Cells; Transcatheter Arterial Chemoembolization; Advanced Liver Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Precision Cells (Experimental): Precision Cells combined with Transcatheter Arterial Chemoembolization:
  Transcatheter Arterial Chemoembolization:
  patients will receive MMC,EADM hepatic arterial infusion,6 cycles. Precision Cells：After accepting concurrent TACE treatment,patients will receive 3 cycles of Precision Cells treatment
  Interventions: Procedure: TACE; Biological: Precision Cells
- Transcatheter Arterial Chemoembolization (Active Comparator): patients will receive MMC,EADM hepatic arterial infusion,6 cycles.
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: TACE — Lipiodol 10-20ml,MMC 8～10mg,EADM20～40mg.According to tumor area of maximum diameter,0.1～0.2ml/cm2 Hepatic arterial infusion.
Biological: Precision Cells — DC cell suspension (1×107 DC+ physiological saline + 0.25% human bloodalbumin) 1ml for each infusion, subcutaneous injection for each infusion 3 cycles, each cycle received two infusions on day 19, 20; 40, 41; 61, 62. Precision cells suspension (1-6×109 Precision cells + physiological saline + 0.25% human bloodalbumin) 300ml for each infusion, IV (in the vein) for each infusion 3 cycles, each cycle received one infusions on day 21, 42, 63.
  Arms: Precision Cells

SUMMARY:
Objectives:

To evaluate the safety and effectiveness of cell therapy using Precision Cells Combined With TACE in Advanced Liver Cancer.

Eligibility:

Individuals greater than or equal to 18 years of age and less than or equal to 65 years of age who have been diagnosed with Advanced Liver Cancer.

DETAILED DESCRIPTION:
A total of 40 patients may be enrolled over a period of 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~65 years old, male or female;
* Life expectancy≥6 months;
* ECOG score: 0-3;
* Advanced Malignancies (lung cancer, gastric cancer) were diagnosed by pathological or clinical physicians,and Diagnosis of hepatocellular carcinoma (HCC), surgery can not be performed but TACE treatment can be carried out;
* Enough venous channel, no other contraindications to the separation and collection of white blood cells;
* Laboratory examination: white blood cell≥3 x 10*9/L, blood platelet count≥60 x 10*/L, hemoglobin≥85g/L; lymphocyte count≥15%, total bilirubin≤100 mol/L; ALT and AST less than five times of the normal level; serum creatinine less than 1.5 times of the normal level;
* Signed informed consent;
* Women of child-bearing age must have evidence of negative pregnancy test and be willing to practice birth control after 2 weeks following the cells transfusion.

Exclusion Criteria:

* Expected Overall survival < 3 months;
* The tumor size or quantity is not suitable for interventional treatment or portal vein tumor thrombus;
* Liver function is Childs Pugh C;
* Had received TACE therapy previously or in radiotherapy at present,or taking Sola Feeney;
* Other serious diseases:the heart,lung, kidney, digestive, nervous, mental disorders, immune regulatory diseases, metabolic diseases, infectious diseases, etc;
* Unable or unwilling to provide informed consent, or fail to comply with the test requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-03 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
Progress-free survival | 2 years

SECONDARY OUTCOMES:
Quality of life | 2 years
  Questionnaire will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Naiyan Han, Study Chair — Shanghai International Medical Center
Locations (1):
- Shanghai International Medical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No